CLINICAL TRIAL: NCT00681967
Title: Conventional Postoperative Radiotherapy (Standard Fractionation) Plus Iressa or Hyperfractionated Radiotherapy Plus Cisplatin and Iressa for Advanced Head & Neck Cancer: A Phase I Pilot Trial
Brief Title: Postoperative Radiotherapy Plus Iressa or Radiotherapy Plus Cisplatin and Iressa for Advanced Head & Neck Cancer
Acronym: IRESSA&H&N
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr. med. Dirk Schneider, AstraZeneca AG Switzerland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0525
Record Dates: First submitted 2008-05-20; First posted 2008-05-21 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Head and Neck Cancer
Keywords: squamous cell cancer of the head & neck; Gefitinib; IRESSA; EGFR Inhibitor; EGFR-tyrosine kinase inhibitor; Subjects with histologically proven squamous cell cancer of the head & neck; Cohort 1:qualifying for postoperative radiotherapy; (pT3, pT4, pN2b, pN2c, pN3).; Cohort 2:qualifying for definite chemoradiotherapy; (Lateral oropharynx, tonsils: T1N2b-3, T2N1-3, T3any N;; Base of tongue, vallecula: T1N1-3, T2-4 any N; Oral cavity,; glottic and supraglottic larynx; Any TN1-3, T3-4 any N;; Hypopharynx: T1N1-3, T2-4 and N)
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): post operative combination of gefinib and RT
  Interventions: Drug: Gefitinib
- Cohort 2 (Experimental): combination of gefitinib with RT and Chemotherapy in non operated patients
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — 250 mg; oral
  Other Names: IRESSA (TM)
  Arms: Cohort 1
Drug: Gefitinib — 250mg; oral
  Other Names: IRESSA (TM)
  Arms: Cohort 2

SUMMARY:
To evaluate the feasibility and safety of (cohort 1) postoperative standard fractionation radiotherapy plus Iressa and of (cohort 2) hyperfractionated radiotherapy plus cisplatin and Iressa

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age over 18 years
* Histologically proven squamous cell cancer of the head & neck (SCCHN)
* Indication for postoperative Radiotherapy: pT3, pT4, pN2b, pN2c, pN3

Exclusion Criteria:

* Hypersensitivity to ZD1839 or any of the excipients of this product
* Tumour stage M1
* Co-existing malignancies diagnosed within the last 5 years. Exceptions: basal cell carcinoma, cervical cancer in situ
* Absolute neutrophil counts <1.5 x 109

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility and safety of (cohort 1) postoperative standard fractionation radiotherapy plus Iressa and of (cohort 2) hyperfractionated radiotherapy plus cisplatin and Iressa

SECONDARY OUTCOMES:
Both cohorts overall survival (OS) local control (LC) rate at six months and at one year
Cohort 1 only time-to-recurrence (TTR)
Cohort 2 only time-to-progression (TTP). Complete Response (CR) rate time to treatment failure (TTF)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Rochlitz, Prof Dr med, Principal Investigator — University Hospital of Basel; Madeleine Billeter, MD, Study Director — AstraZeneca AG, Grafenau 10; 6300 Zug; Switzerland; Verena Renggli, Study Chair — AstraZeneca AG, Grafenau 10; 6300 Zug; Switzerland
Locations (2):
- Switzerland (2):
  - Research Site, Basel
  - Research Site, Bern